CLINICAL TRIAL: NCT02810509
Title: Quality of Anticoagulation With Warfarin in Patient With Atrial Fibrillation for Secondary Stroke Prevention in Korea
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Keun-Sik Hong, Professor, Inje University
Other Study IDs: Warfarin TTR-01
Record Dates: First submitted 2015-12-23; First posted 2016-06-23 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Wafarin; Cardioembolic (CE) stroke; ischemic stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Short-term Warfarin-treated cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  3. TTR evaluable days < 90 days
- Long-term Warfarin-treated cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
  3. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  4. TTR evaluable days ≥ 90 days

SUMMARY:
The current study aims to assess the quality of anticoagulation with warfarin in real world practice of secondary stroke prevention in Korean patients with Atrial fibrillation (AF) and to explore predictors for poor International Normalized Range (INR) control.

DETAILED DESCRIPTION:
* To assess the quality of anticoagulation with warfarin in real world practice of Korea for secondary stroke prevention in patients with AF-related Cardioembolic (CE) stroke 1) who initiated warfarin therapy and treatment at least for more than 7 days of warfarin adjustment period (warfarin-initiated cohort), and 2) who initiated and maintained warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period (long-term warfarin-treated cohort).
* To explore predictors for poor INR control.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the warfarin-initiated cohort

1. Admission due to AF-related ischemic stroke
2. Initiation of warfarin therapy and treatment at least for more than 7 days of warfarin adjustment period
3. For TTR calculation, available consecutive INR values ≥3 after the 7 days of warfarin adjustment

Inclusion criteria for the long-term warfarin-treated cohort

1. Admission due to AF-related ischemic stroke
2. Long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
3. For TTR calculation, available consecutive INR values ≥3 after the 7 days of warfarin adjustment
4. TTR evaluable days ≥ 90 days

Exclusion Criteria:

1. AF with mechanical valve
2. Enrollment in anticoagulation randomized clinical trial
3. Enrollment in studies affecting the target INR range.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who admitted to 16 participating centers due to AF-related ischemic stroke between Jan 1, 2011 and Dec 31, 2012 and started warfarin therapy for secondary stroke prevention will be enrolled in this study. The number of patients is expected to be 2,217 for the warfarin-initiated cohort and 1,057 for the long-term warfarin-treated cohort.
Sampling Method: Probability Sample
Enrollment: 1814 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Sik Hong, MD, Phd, Principal Investigator — Department of Neurology, Ilsan Paik Hospital Inje University
Locations (18):
- South Korea (18):
  - Hallym University College of Medicine, Anyang
  - Dong-A University College of Medicine, Busan
  - Yeungnam University School of Medicine, Daegu
  - Dongguk University Ilsan Hospital, Goyang
  - Chonnam National University Medical School, Gwangju
  - Ilsan Paik Hospital Inje University, Ilsan
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju National University College of Medicine, Jeju City
  - Seoul National University Bundang Hospital, Seongnam
  - Eulji General Hospital, Eulji University School of Medicine, Seoul
  - Korea University College of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul Medical Center, Seoul
  - Seoul National University College of Medicine, Seoul
  - Soonchunhyang University College of Medicine, Seoul
  - Soonchunhyang University, Seoul
  - University of Ulsan College of Medicine, Seoul
  - Yonsei University College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Term Wafarin-treated Cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  3. TTR evaluable days < 90 days
- Long Term Warfarin-treated Cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
  3. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  4. TTR evaluable days ≥ 90 days
Period: Overall Study
Arm/Group | Short Term Wafarin-treated Cohort | Long Term Warfarin-treated Cohort
Started | 584 | 1230
Completed | 584 | 1230
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of Baseline participants are divided by short term and Long term Warfarin-treated cohort.
Groups:
- Long Term Warfarin-treated Cohort: 1. Admission due to AF-related ischemic stroke
  2. Long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
  3. For Time in TTR calculation, available consecutive INR values ≥3 after the 7 days of warfarin adjustment
  4. TTR evaluable days ≥ 90 days
- Total: Total of all reporting groups
Arm/Group | Short Term Wafarin-treated Cohort | Long Term Warfarin-treated Cohort | Total
Number analyzed (Participants) | 584 | 1230 | 1814
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.71 (9.60) | 70.08 (9.73) | 71.25 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 523 | 821
  Male | 286 | 707 | 993

OUTCOME MEASURES:

1. Primary Outcome: Time in TTR, the Percentage of Time in the Therapeutic Range of INR Between 2.0-3.0.
Description: The primary outcome is TTR as measured by the percentage of time in the therapeutic range of INR between 2.0-3.0, using the Rosendaal linear interpolation method.
Time Frame: We will analyze INR data of patients who had AF-related ischemic stroke and were treated with warfarin therapy at least for more than 7 days of warfarin adjustment period. (The INR follow up duration: 1 ~ maximum 3 years)
Measure: Mean (Standard Deviation); unit: percentage of time in therapeutic range
Groups:
- Short-term Cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  3. TTR evaluable days < 90 days
- Long-term Cohort: 1. admission due to AF-related ischemic stroke (known AF or newly detected AF)
  2. long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
  3. for TTR calculation, the number of consecutive INR measurements ≥3 after the 7 days of warfarin adjustment
  4. TTR evaluable days ≥ 90 days
Arm/Group | Short-term Cohort | Long-term Cohort
Number analyzed (Participants) | 584 | 1230
percentage of time in therapeutic range | 43.4 (26.3) | 49.1 (20.8)

2. Secondary Outcome: Percentage of INR Values in the Therapeutic Range of 2.0-3.0: Numbers of INR Values Within the Therapeutic Range by the Total Numbers of INR Measured.
Description: The secondary outcome is the percentage of INR values in the therapeutic range of 2.0-3.0: numbers of INR values within the therapeutic range divided by the total numbers of INR measured.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Number of INR measured
Units Other Than Participants: Number of INR measured
Groups:
- Long-term Cohort: 1. Admission due to AF-related ischemic stroke
  2. Long-term warfarin therapy at least for more than 90 days after the 7 days of warfarin adjustment period
  3. For Time in TTR calculation, available consecutive INR values ≥3 after the 7 days of warfarin adjustment
  4. TTR evaluable days ≥ 90 days
Arm/Group | Short-term Cohort | Long-term Cohort
Number analyzed (Participants) | 584 | 1230
Number analyzed (Number of INR measured) | 8693 | 33941
Number of INR measured | 3900 | 15120

ADVERSE EVENTS:
Time Frame: This is an investigator-initiated study of a retrospective observation study therefore, adverse events and serious adverse events are not collected through this study.
Description: This is an investigator-initiated study of a retrospective observation study therefore, adverse events and serious adverse events are not collected through this study.
Groups:
- Warfarin-initiated Cohort: 1. Admission due to AF-related ischemic stroke
  2. Initiation of warfarin therapy and treatment at least for more than 7 days of warfarin adjustment period
  3. For Time in therapeutic range (TTR) calculation, available consecutive INR values ≥3 after the 7 days of warfarin adjustment
Arm/Group | Warfarin-initiated Cohort | Long Term Warfarin-treated Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No